CLINICAL TRIAL: NCT05482594
Title: Stem Cell Factor, a Potential Biological Marker of Skin Involvement in Systemic Sclerosis?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, BADOT, Valerie, Head of Rhumatology Department, Brugmann University Hospital
Other Study IDs: CHUB-SCF
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Microscopic Angioscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic sclerosis: Patients followed regularly at CHU Brugmann in rheumatology/Dermatology for limited or diffuse systemic sclerosis in accordance with the ACR/EULAR 2013 criteria.
  Interventions: Diagnostic Test: ELISA; Diagnostic Test: Videocapillaroscopy
- Control: Control patients recruited among patients followed for mechanical pathology in rheumatology.
  Interventions: Diagnostic Test: ELISA; Diagnostic Test: Videocapillaroscopy

INTERVENTIONS:
Diagnostic Test: ELISA — During routine blood sampling, serum after centrifugation will be stored and frozen at -80°C in the immunology laboratory in order to carry out analyzes by the ELISA method to measure the levels of SCF.
Diagnostic Test: Videocapillaroscopy — Videocapillaroscopy is a non-invasive and safe method for the morphological examination and the analysis of abnormalities of the microcirculation linked in particular to systemic scleroderma. Here it is a digital capillaroscopy used routinely at the CHU Brugmann, in the follow-up of patients and whose results will be collected in this study.

SUMMARY:
This project aims to study systemic sclerosis and find a serum marker of its cutaneous involvement.

Systemic sclerosis (SSc) is a rare immune disease that is part of connectivitis and is characterized by fibrosis and vasculopathy. Multiple visceral lesions involving these two processes make up the severity of this disease. Its dermatological involvement is a fundamental clinical element.

Systemic sclerosis is mainly divided into two subtypes, depending on the extent of dermatological involvement: limited and diffuse systemic sclerosis. These also differ in certain autoantibody profiles and clinical features. Nevertheless, it is still necessary to determine certain criteria, markers, making it possible to distinguish at an early stage the presence of limited or diffuse systemic sclerosis. The latter being characterized by more severe organic and cutaneous involvement and excess mortality. This would allow for more aggressive management from the outset at an early onset of the disease.

In general, it is known that this pathology is characterized by dysfunction of endothelial cells (EC) and fibroblasts as well as autoimmunity. Many mediators contribute to the fibroblast activation observed in SSc. However, transforming growth factor beta (TGFβ) is considered to be the central regulatory factor of fibrosis processes.

It is also known that endothelial cells interact with mast cells through the production of Stem Cell Factor (SCF) to induce their proliferation and differentiation. The damaged skin tissues in systemic sclerosis are infiltrated in particular by mast cell cells which produce TGFβ.

The team of Kihira et al (1998) demonstrated the presence of a high level of SCF in the serum of patients with systemic sclerosis.

Few studies explore this possible production pathway of TGFβ in systemic sclerosis via SCF assay.

This study will allow the investigators to:

* study this possible route of fibrosis through the dosage of SCF in the serum of patients suffering from systemic sclerosis
* describe SCF as a possible biomarker of skin involvement by hypothesizing that the dosage of SCF will be higher in patients with diffuse scleroderma compared to those with limited scleroderma

ELIGIBILITY:
Inclusion Criteria:

* Patients followed regularly at CHU Brugmann in Rheumatology/Dermatology for limited or diffuse systemic sclerosis in accordance with the ACR/EULAR 2013 criteria.
* Control patients recruited among patients followed for mechanical pathology in rheumatology

Exclusion Criteria:

* Patients with comorbidities of hematological diseases, asthma or severe chronic renal failure (GFR < 30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed regularly at CHU Brugmann in Rheumatology/Dermatology for limited or diffuse systemic sclerosis in accordance with the ACR/EULAR 2013 criteria.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Stem Cell Factor | 1 year
  Stem Cell Factor blood levels
Videocapillaroscopy imaging report | 1 year
  Videocapillaroscopy is a non-invasive and safe method for the morphological examination and the analysis of abnormalities of the microcirculation linked in particular to systemic scleroderma.

CONTACTS AND LOCATIONS:
Overall Officials: WEYNAND Marjolaine, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No